CLINICAL TRIAL: NCT04198818
Title: A First-in-Human, Open Label, Phase I/II Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HH2710 in Patients With Advanced Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HH2710 in Patient With Advanced Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor business decision
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH2710-G101
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Advanced Tumors; Melanoma; Non-Small-Cell Lung Cancer; Erdheim-Chester Disease; Other RAS/RAF/MEK/ERK Mutated Tumors
Keywords: Melanoma; Non-Small-Cell Lung Cancer; Erdheim-Chester Disease; MAPK pathway; ERK1; ERK2
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Erdheim-Chester Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation study of HH2710 (Experimental): to determine the MTD of HH2710 and/or Recommended Phase II dose (RP2D).
  Interventions: Drug: HH2710

INTERVENTIONS:
Drug: HH2710 — HH2710 is a small molecule that potently inhibits both ERK1 and ERK2 protein kinases in the nanomolar range. The kinase selectivity assessment towards a panel of over 400 protein kinases showed that HH2710 barely inhibited other kinases at a concentration up to 1 μM, except the substantial inhibition against ERK1 (MAPK1), ERK2 (MAPK2) and the MAPK pathway upstream kinases MEK and RAF proteins.

SUMMARY:
This is a First-in-Human, Open Label, Phase I/II Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HH2710 in Patients with Advanced Tumors, composed of a Phase I dose escalation and dose expansion stage and a Phase II dose extension stage.

DETAILED DESCRIPTION:
HH2710 is developed by Shanghai Haihe Pharmaceutical Co., Ltd. HH2710 is a highly potent, selective, reversible, ATP-competitive ERK1/2 inhibitor. This is a first-in-human study of HH2710 and is designed as an open-label, multicenter, Phase I/II study which is composed of a Phase I dose escalation and dose expansion stage and a Phase II dose extension stage.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent prior to initiation of any study-related procedures.
2. Male or female patients aged ≥ 18 years.
3. Phase I dose escalation stage: Patients who have been diagnosed with histologically or cytological documented, unresectable/metastatic tumors that are refractory or intolerant to standard therapy or for whom no curative standard therapy exists.

   - For LCH/ECD: Eligible patients must have multifocal disease and the diagnosis must be confirmed by pathological evaluation of the affected tissue.
4. Phase I expansion stage and Phase II stage: Histologically or cytologically documented unresectable/metastatic tumors with evidence of genetic mutations affecting MAPK pathway is required. Patients with a BRAF V600 mutation must have progressed on or after standard therapy, including BRAF and/or MEK inhibitors (≤3 lines). Patients entering the Phase 2 portion of the trial will be enrolled in Cohorts 1-4 depending upon their tumor type.

   * Cohort 1: Patients with BRAF/NRAS (mutation sites as follows: NRAS G13V, NRAS Q61, BRAF V600, BRAF G469A, L485W, L597Q, T599dup) mutated melanoma;
   * Cohort 2: Patients with BRAF/NRAS (mutation sites as follows: NRAS G13V, NRAS Q61, BRAF V600, BRAF G469A, L485W, L597Q, T599dup) mutated non-small cell lung cancer;
   * Cohort 3: Patients with BRAF V600 mutated Langerhans Cell Histiocytosis Syndrome (LCH)/ Erdheim-Chester disease (ECD);
   * For LCH/ECD: Eligible patients must have multifocal disease and the diagnosis must be confirmed by pathological evaluation of the affected tissue.
   * Cohort 4: Patients with RAS/RAF/MEK/ERK mutated tumor types that are not included in other cohorts.
5. Patients in the Phase I dose escalation portion of the trial may have measurable (per RECIST v1.1) or evaluable disease. Patients in the Phase I expansion and Phase II portions of the trial must have measurable disease per RECIST v1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status≤1.
7. Predicted life expectancy ≥ 3 months;
8. Adequate renal function defined as a creatinine clearance ≥ 60 mL/min;
9. Adequate hepatic function [total bilirubin ≤ 1.5 x UNL; AST (aspartate aminotransferase) and ALT (alanine aminotransferase) ≤ 3 x UNL or ≤ 5 x UNL if due to liver involvement by tumor];
10. Adequate cardiac function, > institutional lower limit of normal e.g., left ventricular ejection fraction (LVEF) of ≥ 50% as assessed by ultrasound/echocardiography (ECHO) or multi-gated acquisition (MUGA) ; corrected QT interval (QTcF) < 460 ms (male patients), < 470 ms (female patients) (using QTc Fridericia's formula.
11. Adequate bone marrow function, patients must not have required blood transfusion or growth factor support ≤ 7 days before sample collection for the following ：

    • Absolute neutrophil count ≥ 1.5 × 109/L; • Hemoglobin ≥ 9 g/dL; • Platelet count ≥100 × 109/L; • International normalized ratio (INR) ≤ 1.5; • Activated partial prothrombin time (APTT) ≤ 1.5 × ULN;
12. Willing and able to participate in the trial and comply with all study requirements;

Exclusion Criteria:

1. Gastrointestinal condition which could impair absorption of study medication;
2. Congenital long QT syndrome, or any known history of torsade de pointes (TdP), or family history of unexplained sudden death;
3. Clinically uncontrolled hypertension (after standard antihypertensive treatment, systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg);
4. Undergone a bone marrow or solid organ transplant;
5. Any toxicities from prior treatment that have not recovered to ≤ CTCAE Grade 1 before the start of study drug, with the exception of hair loss or fatigue;
6. Patients who have previously participated in clinical trials of ERK inhibitors drug;
7. Allergic to similar drugs or their excipients;
8. HIV (human immunodeficiency virus) infection, active hepatitis B or hepatitis C patients (HBsAg positive patients also detected HBV (hepatitis B virus) DNA ≥ 103 copies or ≥ 200 IU/ml; HCV antibody test results are positive, and HCV (hepatitis C virus) RNA PCR test results are positive);
9. Uncontrolled or severe intercurrent medical condition:

   * Unstable angina pectoris ≤3 months prior to starting study drug;
   * Acute myocardial infarction ≤3 months prior to starting study drug;
10. Symptomatic CNS metastases that are neurologically unstable or requiring increasing doses of steroids to control CNS disease. Note: Controlled CNS metastases are allowed. Radiotherapy or surgery for CNS metastases must have been completed >2 weeks prior to study entry. No new neurologic deficits on clinical examination and no new findings on CNS imaging are permitted. Steroid use for management of CNS metastases must be at a stable dose for two weeks preceding study entry;
11. Any cancer-directed therapy (chemotherapy, radiotherapy, hormonal therapy, biologic or immunotherapy, Chinese medicine/Chinese patent medicine with anti-tumor effect, etc.) within 28 days or 5 half-lives, whichever is shorter;
12. Major surgery within 4 weeks prior to first dose;
13. Any use of an investigational drug within 28 days or 5 half-lives (whichever is shorter) prior to the first dose of HH2710;
14. Pregnant or breast-feeding women;
15. Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc.

    * Severe infections within 4 weeks prior to the first dose, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
    * Received therapeutic oral or IV antibiotics within 2 weeks prior to the first dose of study drug.
16. Any important or severe medical illness or abnormal laboratory finding that would increase the risk of participating in this study;
17. A history or current evidence/risk of retinal vein occlusion, central serous retinopathy or choroidneovascularization (CNV) ;
18. Concurrent therapy with any other investigational agent;
19. Concomitant malignancies or previous malignancies with less than 2 years disease-free interval at the time of enrollment; (But basal cell carcinoma skin cancer, cervical CIS(carcinoma in situ), CIS of the breast, localized or low Gleason grade prostate cancer, and < T2 bladder cancer can be included);
20. Current treatment with agents including vitamins, supplements, and herbal supplements that are metabolized solely through CYP3A4;
21. Severe chronic obstructive pulmonary disease, severe asthma, pneumoconiosis, asbestosis and other occupational lung diseases.
22. A history of acute or chronic pancreatitis, surgery of the pancreas, or any risk factors that may increase the risk of pancreatitis;
23. Contraception: Patients who do not meet the following conditions will be excluded, - For women: Negative pregnancy test for females of child-bearing potential; must be surgically sterile, postmenopausal (defined as no menstrual cycle for at least 12 consecutive months), or compliant with an acceptable contraceptive regimen (2 highly effective forms, such as oral contraceptives, condom with spermicide, etc.) during and for 6 months after the treatment period. Abstinence is not considered an adequate contraceptive regimen; - For men: Must be surgically sterile, or compliant with a contraceptive regimen (as above) during and for a minimum of 6 months after the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Horizon Oncology Research, LLC, Lafayette, Indiana
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
- Shanghai East hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HH2710 25mg BID: administered orally，25mg QD at C1D1, then 25mg BID from C1D2 (21 days/cycle).
- HH2710 50mg BID: administered orally，50mg BID (21 days/cycle)
- HH2710 100mg BID: administered orally，100mg BID(21 days/cycle)。
- HH2710 300mg QD: administered orally，300mg QD (21 days/cycle)
- HH2710 400mg QD: administered orally，400mg QD (21 days/cycle)
- HH2710 600mg QD: administered orally，600mg QD (21 days/cycle)
- HH2710 800mg QD: administered orally，800mg QD (21 days/cycle)
- HH2710 200mg BID: administered orally，200mg BID (21 days/cycle)
Period: 25mg BID
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD | HH2710 200mg BID
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 50mg BID
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD | HH2710 200mg BID
Started | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Period: 100mg BID
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD | HH2710 200mg BID
Started | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Period: 300mg QD
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD | HH2710 200mg BID
Started | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Period: 400mg QD
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD | HH2710 200mg BID
Started | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Period: 600mg QD
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD | HH2710 200mg BID
Started | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0
Period: 800mg QD
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD | HH2710 200mg BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Period: 200mg BID
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD | HH2710 200mg BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- HH2710 25mg BID: administered orally，25mg QD at C1D1, then 25mg BID from C1D2 (21 days/cycle.
- HH2710 200mg BID: administered orally，200mg BID(21 days/cycle)。
- Total: Total of all reporting groups
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD | Total
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 4 | 4 | 8 | 4 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 5 | 4 | 2 | 5 | 2 | 26
  >=65 years | 0 | 1 | 1 | 2 | 0 | 2 | 3 | 2 | 11
Age, Continuous [Median (Full Range); unit: years] | 53 [53 to 57] | 51 [45 to 78] | 55 [43 to 75] | 57 [37 to 77] | 55 [39 to 63] | 63 [35 to 71] | 62 [29 to 76] | 54 [39 to 70] | 57 [29 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 4 | 3 | 3 | 4 | 1 | 19
  Male | 1 | 3 | 2 | 3 | 1 | 1 | 4 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 4 | 7 | 4 | 4 | 7 | 4 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 7 | 0 | 1 | 5 | 2 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 5
  White | 1 | 2 | 2 | 0 | 2 | 3 | 2 | 2 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Median (Full Range); unit: cm] | 170.10 [165.1 to 183.0] | 173.40 [170.3 to 179.0] | 173.30 [167.4 to 177.8] | 161.40 [155.0 to 175.0] | 168.05 [162.5 to 175.9] | 161.90 [156.8 to 172.7] | 167.50 [155.0 to 183.2] | 167.75 [143.0 to 198.6] | 167.40 [143.0 to 198.6]
Weight [Mean (Standard Deviation); unit: kg] | 78.97 (24.568) | 68.83 (12.744) | 78.75 (13.550) | 65.29 (7.370) | 88.30 (23.527) | 65.15 (17.241) | 69.21 (17.960) | 74.38 (20.852) | 72.44 (17.098)
BMI [Median (Standard Deviation); unit: kg/m2] | 26.57 (8.693) | 22.80 (5.237) | 26.38 (4.597) | 24.80 (2.749) | 31.58 (10.449) | 24.53 (6.856) | 24.20 (5.182) | 25.58 (1.193) | 25.61 (5.705)
ECOG Performance Status [Count of Participants; unit: Participants] — Inclusion criteria 6. Eastern Cooperative Oncology Group (ECOG) performance status≤ 1. And 0 is better than 1.
  Grade 0 means Asymptomatic, fully active, able to carry on all pre-disease activities without restriction.
  Grade 1 means Symptomatic but completely ambulatory, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work.
  Participants
    0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 6
    1 | 2 | 3 | 3 | 7 | 4 | 3 | 6 | 3 | 31
Tumor Histology type, n (%) [Count of Participants; unit: Participants]
  Adenocarcinoma | 2 | 3 | 1 | 5 | 4 | 3 | 4 | 3 | 25
  Carcinoid Carcinoid Carcinoid | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Endometrioid | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Invasive Ductal Carcinoma | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 4
  Melanoma | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Squamous Cell Carcinoma | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  other | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Tumor Current Stage, n (%) [Count of Participants; unit: Participants] — Tumor stage is decided by the clinical diagnose of the investigator according to the treatment guideline of the particular tumor type. Generally,Stage I: The tumor is small and contained within the organ it started in. Stage II: tumor is larger but not spread into the surrounding tissues. Stage III: tumor spread into surrounding tissues. Stage IV: tumor has spread to another body organ. Generally,stage I is better than stage II. A and B is subgrade of each stage, and A generally means tumor size is smaller than B.
  Participants
    Stage III | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Stage IIIB | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Stage IV | 3 | 1 | 3 | 6 | 3 | 4 | 7 | 4 | 31
    Stage IVA | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
    Unknown | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Location of metastases at baseline [Number; unit: sites]
  Adrenal | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Axillary Lymph Nodes | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 5
  Bladder | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Bone | 1 | 1 | 1 | 2 | 0 | 1 | 3 | 1 | 10
  Bone, Lumbar Vertebrae | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Bone, Sacrum | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Brain | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3
  Cervical Lymph Node | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 4
  Colon | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Kidney | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
  Liver | 3 | 2 | 2 | 4 | 4 | 3 | 5 | 3 | 26
  Lung | 0 | 3 | 2 | 5 | 3 | 1 | 7 | 4 | 25
  Meninges | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Omentum | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Pancreas | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Pericardial Effusion (Malignant) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Peritoneum | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 5
  Pleura | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 4
  Pleural Effusion (Malignant) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Spleen | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Stomach | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Thoracic Lymph Nodes | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Other | 3 | 2 | 4 | 6 | 1 | 2 | 3 | 3 | 24
Number of metastases at baseline [Count of Participants; unit: Participants]
  1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 6
  2 | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 7
  3 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 6
  >3 | 1 | 1 | 1 | 1 | 0 | 1 | 6 | 2 | 13
  Missing | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 5
Number of prior lines or regimens of therapy [Number; unit: number of lines or regimens]
  First Line | 2 | 2 | 3 | 6 | 2 | 3 | 7 | 1 | 26
  Second Line | 2 | 2 | 3 | 6 | 2 | 3 | 5 | 0 | 23
  Third Line | 2 | 2 | 3 | 3 | 1 | 3 | 4 | 1 | 19
  Third Line More | 1 | 2 | 3 | 2 | 1 | 2 | 3 | 0 | 14
  Neo-adjuvant | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Adjuvant | 0 | 0 | 0 | 3 | 1 | 0 | 3 | 1 | 8
  Palliative | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Other | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: MTD (Maximum Tolerated Dose)
Description: MTD estimation: After the escalation is completed, select the MTD based on the isotonic regression. Specifically, select the MTD for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate. If there are ties, select the higher dose level when the isotonic estimate is lower than the target toxicity rate and select the lower dose level when the isotonic estimate is greater than or equal to the target toxicity rate.
Time Frame: Up to 1 cycle (21 days)
Measure: Number; unit: mg
Groups:
- All Participants: All participants received at least one dose of the study treatment.
Arm/Group | All Participants
Number analyzed (Participants) | 37
mg | NA — Insufficient number of participants with events because of the early termination of the study.

2. Primary Outcome: Number of Participants Who Experienced DLT (Dose Limiting Toxicities)
Description: DLT is defined as: any toxicity meeting the specified criteria and considered at least possibly related to HH2710 (i.e., any toxicity for which a clear alternative etiology such as disease progression has not been identified) should be considered a DLT per National Cancer Institute Common Terminology Criteria for Adverse events (NCI-CTCAE V5.0) standard, which met any of the following, NCI-CTCAE V5.0 will be used for all grading, and compliance of 80% (i.e. 17 of 21 days) in Cycle 1 is required for a patient to be included in the DLT evaluation. For the purpose of dose-escalation decisions, DLTs will be considered and included in the BOIN.
Time Frame: Up to 1 cycle (21 days)
Measure: Count of Participants; unit: Participants
Groups:
- HH2710 100mg BID: administered orally，100mg BID(21 days/cycle)
- HH2710 200mg BID: administered orally，200mg BID(21 days/cycle)
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 4 | 4 | 8 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

3. Primary Outcome: Tumor Objective Response Rate (ORR)
Description: ORR=CR+PR. ORR was defined as the percentage of patients who had at least one confirmed response of CR or PR defined by RECIST version 1.1 prior to any evidence of progression, and was calculated and summarized by the treatment group, along with the 95% confidence interval (CI) calculated by the Clopper-Pearson method.
Time Frame: Up to 1 cycle (21 days)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 4 | 4 | 8 | 4
percentage of patients | 0 [0 to 70.8] | 0 [0 to 70.8] | 0 [0 to 60.2] | 0 [0 to 41.0] | 0 [0 to 60.2] | 0 [0 to 60.2] | 0 [0 to 36.9] | 0 [0 to 60.2]

4. Secondary Outcome: Pharmacokinetic Measures - Peak Time (Tmax)
Description: Measure of time to reach maximum (peak) plasma concentration(s)
Time Frame: C1D1,pre-dose,15min,30min,1h,2h,3h,4h,6h,8h,12h;C1D2, pre-dose and 24h; C1D7,C1D10, pre-dose.C1D15 at pre-dose,15min,30min,1h,2h,3h,4h,6h,8h,12h, C1D16 pre-dose and 24h,C1D22 pre-dose,and C2D1,C3D1,C5D1,C7D1,C9D1 pre-dose.
Population: Pharmacokinetic data of HH2710 following a single and multiple dosing administration was evaluated in 35 and 25 patients, respectively.All patients received at least one dose of the study treatment and were included in the FAS and SAS. 35 patients were included in PKS. and group analysis is based on dose administration group.
Measure: Mean (Full Range); unit: h
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 3 | 4 | 7 | 4
h
  Single Dose Administration | 1 [0.5 to 3] | 2 [1 to 2] | 2.5 [1 to 24] | 2 [1 to 24] | 4 [1 to 24] | 2.5 [2 to 3] | 2 [0.5 to 4] | 7 [3 to 8]
  Multiple-dose Administration: number analyzed (Participants) | 3 | 2 | 4 | 3 | 3 | 4 | 6 | 0
  Multiple-dose Administration | 1 [1 to 24] | 1.5 [1 to 2] | 2 [2 to 2] | 3 [2 to 3] | 8 [1 to 24] | 6 [2 to 8] | 4 [2 to 24] |

5. Secondary Outcome: Pharmacokinetic Measures - Peak Plasma Concentration (Cmax)
Description: Measure the maximum (peak) plasma concentration(s)
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 3 | 4 | 7 | 4
ng/mL
  Single Dose Administration | 281 (37.1) | 382 (59.7) | 826 (66.1) | 1440 (70.2) | 1389 (131.1) | 1926 (82.5) | 3462 (45.6) | 5313 (88.0)
  Multiple-dose Administration: number analyzed (Participants) | 3 | 2 | 4 | 3 | 3 | 4 | 6 | 0
  Multiple-dose Administration | 920 (77.2) | 1038 (22.0) | 2115 (17.1) | 2130 (61.2) | 1112 (42.6) | 1933 (83.3) | 6519 (6519) |

6. Secondary Outcome: Pharmacokinetic Measures - Plasma Concentration Timecurve From Time 0 to Time (t) (AUC0-t)
Description: Measure the variation of concentration in blood plasma as a function of time
Time Frame: as for outcome 4
Population: Pharmacokinetic data of HH2710 following a single and multiple dosing administration was evaluated in 35 and 25 participates, respectively. But the AUC0-t, t1/2, Lambda z (λz) and CL/F of some patients could not be calculated because of insufficient sampling time points after Tmax point during the elimination phase. So the participates analyzed for AUC0-t, t1/2, Lambda z (λz) and CL/F is less than participates of dosing administration.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD
Number analyzed (Participants) | 3 | 3 | 4 | 7 | 3 | 4 | 4 | 4
h*ng/mL
  Single Dose Administration | 2858 (58.4) | 3139 (52.6) | 7683 (61.0) | 16027 (67.0) | 11369 (87.9) | 20546 (66.7) | 37032 (25.8) | 79134 (64.0)
  Multiple-dose Administration: number analyzed (Participants) | 3 | 1 | 4 | 3 | 3 | 4 | 3 | 0
  Multiple-dose Administration | 16619 (108.2) | 13738 (NA) — 1 data so no SD. | 34387 (23.5) | 29611 (91.5) | 17572 (39.6) | 28267 (69.8) | 64857 (95.3) |

7. Secondary Outcome: Pharmacokinetic Measures -Plasma Elimination Half-life (t1/2)
Description: Terminal half-life, defined as 0.693 (ln2) divided by Lambda z. And t1/2，Lambda z (λz), Vz/F, are only applicable for single dose administration.
Time Frame: Single dose, C1D1,pre-dose,15min,30min,1h,2h,3h,4h,6h,8h,12h(if available),C1D2, pre-dose(if available)
Population: AUC0-t, t1/2, Lambda z and CL/F of some patients could not be calculated because of insufficient sampling time points after Tmax point during the elimination phase. So the participates analyzed for AUC0-t, t1/2, Lambda z (λz) and CL/F is less than participates of dosing administration.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 4 | 4 | 2
h | 16 (12) | 15.6 (12.6) | 12.2 (6.5) | 37.9 (16.7) | 8.8 (1.1) | 12.4 (3.5) | 8.9 (2.9) | 20.9 (1.1)

8. Secondary Outcome: Pharmacokinetic Measures - Plasma Clearance Rate Constant, Lambda z (λz)
Description: Terminal phase rate constant, determined by linear regression of at least 3 points on the terminal phase of the log-linear plasma concentration-time curve. The correlation coefficient (r2) for the goodness of the fit of the regression line through the data points has to be 0.85 or higher for the value to be considered reliable. If the WinNonlin data points are not on the linear portion of the terminal slope, the data points will be selected manually prior to calculation of Lambda_z.
  And t1/2，Lambda z (λz), Vz/F，these 3 PK parameters are only applicable for single dose administration.
Time Frame: Single dose, C1D1,pre-dose,15min,30min,1h,2h,3h,4h,6h,8h,12h(if available),C1D2, pre-dose(if available)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 4 | 4 | 2
1/h | 6.1 (3.7) | 6.4 (3.7) | 3 (2.6) | 2.2 (1.2) | 8 (1) | 6 (1.6) | 5.4 (3.7) | 3.3 (0.2)

9. Secondary Outcome: Pharmacokinetic Measures - Apparent Clearance (CL/F)
Description: Measure apparent total clearance(s) from plasma after oral
Time Frame: C1D1,pre-dose,15min,30min,1h,2h,3h,4h,6h,8h,12h ;C1D2, pre-dose and 24h; C1D7,C1D10, pre-dose.C1D15 at pre-dose,15min,30min,1h,2h,3h,4h,6h,8h,12h, C1D16 pre-dose and 24h,C1D22 pre-dose,and C2D1,C3D1,C5D1,C7D1,C9D1 pre-dose.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 4 | 4 | 2
L/h
  Single Dose Administration: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 4 | 4 | 2
  Single Dose Administration | 8.2 (5.6) | 14.7 (9.5) | 9.3 (4.7) | 13.6 (19.3) | 26.5 (21.2) | 23.3 (21.6) | 14.4 (5) | 4.1 (1.6)
  Multiple-dose Administration: number analyzed (Participants) | 3 | 2 | 4 | 3 | 3 | 4 | 2 | 0
  Multiple-dose Administration | 5.1 (3.2) | 5.9 (0.1) | 5.5 (1.2) | 21.3 (18.8) | 18.9 (7) | 18.5 (8.7) | 6.8 (2.8) |

10. Secondary Outcome: Pharmacokinetic Measures - Apparent Volume of Distribution (Vz/F)
Description: The apparent volume of distribution during terminal phase (associated with λz)(volume). And t1/2，Lambda z (λz), Vz/F，these 3 PK parameters are only applicable for single dose administration.
Time Frame: Single dose, C1D1,pre-dose,15min,30min,1h,2h,3h,4h,6h,8h,12h(if available),C1D2, pre-dose(if available)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 4 | 4 | 2
L | 126.5 (30.4) | 218.9 (32.3) | 151.9 (104.7) | 454 (505) | 353 (311.6) | 385 (328) | 184 (82) | 122 (42)

ADVERSE EVENTS:
Time Frame: up to 30 days after the last dose administration for each participate, and an average of 24 weeks.
Arm/Group | HH2710 25mg BID | HH2710 50mg BID | HH2710 100mg BID | HH2710 200mg BID | HH2710 300mg QD | HH2710 400mg QD | HH2710 600mg QD | HH2710 800mg QD
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3 | 1/4 | 4/7 | 1/4 | 2/4 | 6/8 | 2/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/4 | 3/7 | 3/4 | 1/4 | 5/8 | 1/4
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 4/4 | 7/7 | 4/4 | 4/4 | 8/8 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HH2710 25mg BID (N=3) | HH2710 50mg BID (N=3) | HH2710 100mg BID (N=4) | HH2710 200mg BID (N=7) | HH2710 300mg QD (N=4) | HH2710 400mg QD (N=4) | HH2710 600mg QD (N=8) | HH2710 800mg QD (N=4)
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Central serous chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystoid macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HH2710 25mg BID (N=3) | HH2710 50mg BID (N=3) | HH2710 100mg BID (N=4) | HH2710 200mg BID (N=7) | HH2710 300mg QD (N=4) | HH2710 400mg QD (N=4) | HH2710 600mg QD (N=8) | HH2710 800mg QD (N=4)
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 6 | 1 | 2 | 3 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 3 | 1 | 2 | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3 | 1 | 1 | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 4 | 2 | 1 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 0 | 2 | 4 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 2 | 0 | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 3 | 1 | 1 | 3 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT04198818/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT04198818/SAP_001.pdf
  • Informed Consent Form (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04198818/ICF_002.pdf